CLINICAL TRIAL: NCT04284241
Title: Parents' Health-Education Handbook in Preventing Pediatric Urolithiasis in Kashgar Region of China: A Clustered Randomized Controlled Trial
Brief Title: Parents' Health-Education Handbook in Preventing Pediatric Urolithiasis Formation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guohua Zeng (Other)
Responsible Party: Sponsor-Investigator, Guohua Zeng, Vice-president, The First Affiliated Hospital of Guangzhou Medical University
Organization: The First Affiliated Hospital of Guangzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MRER(72)2017
Record Dates: First submitted 2018-10-21; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Urolithiasis
Keywords: Pediatric urolithiasis; Uyghur; Parents'Health-Education Handbook
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants include newborns and their parents. The baseline of newborns includes demographic data, blood cell analysis, urinary tract ultrasonographic examination. Parents will be asked to answer a questionnaire which regarding the knowledge, attitudes, and practices (KAP questionnaire) related to pediatric stone. Parents also undergo and active health education by the investigator with the " Parents' Health-Education Handbook", and Handbook will be given to them. Handbook includes the knowledge of symptoms, hazards, epidemiology, risk factors, therapy, and prevention of pediatric urolithiasis, and also baby's right feeding methods. Follow up is made every year in the first three years, and the program is done as the baseline.
  Interventions: Behavioral: Parents'Health-Education Handbook
- Control group (No Intervention): Participants include newborns and their parents. The baseline of newborns includes demographic data, blood cell analysis, urinary tract ultrasonographic examination. Newborns' parents will be asked to answer a questionnaire which regarding the knowledge, attitudes, and practices (KAP questionnaire) related to pediatric stone. But parents do not undergo active health education. And Handbook will not be given to them. However, a poster which has the same content as the Handbook is normally displayed in the maternity ward. Parents have the opportunity to see the poster, but without any special remind. Follow up is made every year in the first three years, and the program is done as the baseline.

INTERVENTIONS:
Behavioral: Parents'Health-Education Handbook — We created a Parents' Health-Education Handbook to teach the newborns' parents to enhance their knowledge of pediatric stone, with a view to changing parents' cognition, attitude and behavior for preventing pediatric stone formation by this cluster randomized control trail.
  Arms: Intervention group

SUMMARY:
The aim of this study is to estimate the role of Parents' Health-Education Handbook in preventing pediatric urolithiasis. This study is designed as an unmatched clusters randomized intervention trial. A total of 171 villages and communities in Shufu Count in Kashgar Region of China are assigned to intervention group or control group by a simple random sampling technique with a rate of 1:1. Newborns and their parents are assigned to intervention group or control group as their villages or communities. And at least 2314 newborns are needed in this study. Participants include newborns and their parents. The baseline of newborns includes demographic data, blood cell analysis, urinary tract ultrasonographic examination. Newborns' parents will be asked to answer a questionnaire which regarding the knowledge, attitudes, and practices (KAP questionnaire, estimated by scores) related to pediatric stone. Parents in intervention group will undergo and active health education by the investigator with " Parents' Health-Education Handbook", while parents in control group are without the program. Newborns are invited to undergo blood cell analysis, urine analysis and urinary tract ultrasonographic examination separately when they are one, two and three years old. Their parents will be asked to answer the same KAP questionnaire at the same time. The incidence of urolithiasis is evaluated and compared between the two groups. Improvement of knowledge, attitudes, and practices (KAP questionnaire) related to pediatric stone of parents are evaluated. Association between urolithiasis incidence and improvement of scores in KAP questionnaire are evaluated.

DETAILED DESCRIPTION:
Pediatric urolithiasis is a very common disease among Uyghur children of China. Investigators have conducted a cross-sectional survey among children≤14 years in Kashgar Region, which is Uyghur concentrated region and lies in southern Xinjiang Uyghur Autonomous Region July to December 2016. The results showed that the current prevalence rate of urolithiasis was 1.8% among children ≤14 years, while the overall prevalence was 3.6%. The prevalence of urolithiasis for children ≤1 year was 5.63%. Binary logistic regression analysis showed that non-breastfeeding, urinary tract infection, with a family history of urolithiasis and excessive sweating were all statistical significantly associated with increased risk of urinary stone.

Since most of the risks of urolithiasis among Uyghur children are associated with feeding and living habits, investigators create a Parents' Health-Education Handbook based on these results. This Handbook includes the knowledge of symptoms, hazards, epidemiology, risk factors, therapy, and prevention of pediatric urolithiasis, and also baby's right feeding methods. Investigators use this Handbook to teach newborn's parents to enhance their knowledge of pediatric stone, with a view to change parents' cognition, attitude and behavior of preventing stone formation.

This study is designed as an unmatched clusters randomized intervention trial. The aim of this study is to investigate the role of Parents' Health-Education Handbook in preventing pediatric urolithiasis formation. It is conducted in Shufu Count in Kashgar Region of China, which include 171 villages and communities. Investigators define each village or community as a cluster. And these villages and communities are assigned to intervention group or control group by a simple random sampling technique with a rate of 1:1. A total of 86 villages and communities are assigned to intervention group, while 85 villages and communities are assigned to control group. Participants include newborns and their parents. The newborns and their parents are assigned to intervention group or control group as their villages or communities.

The incidence (same as prevalence) of urolithiasis was 5.63% for children ≤1 year by our former study. The intervention (Parents' Health Education) is considered effective when the incidence decreases more than one half (2.8%) for children when they are 1-year old in this study. So for sample size, we estimate the normal incidence of urolithiasis (π0) is about 5.6% , the incidence will decrease to less than 2.8%(π1) after one year intervention, with α of 0.05, 1-β=90%, 1052 newborns are required by the formula for each group; considered a predicted of 10% missed follow-up late, and at least 2314 newborns needed in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Full-term newborn (37-42 weeks pregnant) .
2. The weight is ≥2.5 kg at birth.

Exclusion Criteria:

1. Urinary system congenital malformation.
2. Sponge kidney.
3. Hydronephrosis.
4. Ureteropelvic junction obstruction.
5. Hypospadias.
6. Urinary calculi.
7. congenital heart disease.
8. Down syndrome

Ages: 1 Day to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2500 (Estimated)
Dates: Start 2017-11-20 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of pediatric urolithiasis for the first year. | One year after the child was born.
  When kids are one year old, they will be invited to undergo blood cell analysis, urine analysis and urinary tract ultrasonographic examination separately. If stone is found by ultrasound, low dose urinary CT scan is invited to done. Their parents will be asked to answer the same KAP questionnaire as baseline each time. The incidence of urolithiasis is evaluated and compared between intervention and control groups. Improvement (estimated by scores in KAP questionnaire) of knowledge, attitudes, and practice related to pediatric stone of parents are estimated and compared between two groups. Association between urolithiasis incidence and improvement of scores in KAP questionnaire are evaluated.
The incidence of pediatric urolithiasis for the second year. | Two years after the child was born.
  When kids are two years old, they will be invited to undergo blood cell analysis, urine analysis and urinary tract ultrasonographic examination separately. If stone is found by ultrasound, low dose urinary CT scan is invited to done. Their parents will be asked to answer the same KAP questionnaire as former. The incidence of urolithiasis is evaluated and compared between intervention and control groups. Improvement (estimated by scores in KAP questionnaire) of knowledge, attitudes, and practice related to pediatric stone of parents are estimated and compared between two groups. Association between urolithiasis incidence and improvement of scores in KAP questionnaire are evaluated.
The incidence of pediatric urolithiasis for the third year. | Three years after the child was born.
  When kids are three years old, they will be invited to undergo blood cell analysis, urine analysis and urinary tract ultrasonographic examination separately. If stone is found by ultrasound, low dose urinary CT scan is invited to done. Their parents will be asked to answer the same KAP questionnaire as former. The incidence of urolithiasis is evaluated and compared between intervention and control groups. Improvement (estimated by scores in KAP questionnaire) of knowledge, attitudes, and practice related to pediatric stone of parents are estimated and compared between two groups. Association between urolithiasis incidence and improvement of scores in KAP questionnaire are evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Guohua Zeng, PhD, Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- epartment of Urology, Minimally Invasive Surgery Center, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided